CLINICAL TRIAL: NCT03096743
Title: Evaluating Raised Intracranial Pressure Using MR Elastography
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, John J Chen, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-007037; 5U10EY025990-02 (NIH)
Record Dates: First submitted 2016-12-15; First posted 2017-03-30 (Actual); Last update posted 2025-03-31 (Actual); Status verified 2025-03

CONDITIONS: Idiopathic Intracranial Hypertension
MeSH Terms: conditions — Pseudotumor Cerebri | interventions — Spinal Puncture; Tomography, Optical Coherence; Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Patients with increased intracranial hypertension (Experimental): Patients will receive the MR elastography, MRI structural brain imaging, Optical Coherence Tomography (OCT) imaging, Optic nerve B-scan ultrasound and Lumbar puncture.
  Interventions: Diagnostic Test: MR elastography; Diagnostic Test: MRI structural brain imaging; Procedure: Lumbar puncture; Diagnostic Test: Optical Coherence Tomography (OCT) imaging; Diagnostic Test: Optic nerve B-scan ultrasound
- Patient without raised intracranial hypertension (Experimental): Patients will receive the MR elastography, MRI structural brain imaging, Optical Coherence Tomography (OCT) imaging, and Optic nerve B-scan ultrasound. Some patients will receive lumbar punctures.
  Interventions: Diagnostic Test: MR elastography; Diagnostic Test: MRI structural brain imaging; Diagnostic Test: Optical Coherence Tomography (OCT) imaging; Diagnostic Test: Optic nerve B-scan ultrasound

INTERVENTIONS:
Diagnostic Test: MR elastography — MR elastography image acquisition will be conducted on the Compact 3T MRI scanner using a modified single-shot spin-echo echo-planar imaging pulse sequence.
Diagnostic Test: MRI structural brain imaging — MRI structural brain imaging will be done on the Compact 3T MRI at the same time as MR elastography.
Procedure: Lumbar puncture — All patients with papilledema will get lumbar punctures with opening pressure as part of their work-up for papilledema. A small number of patients without increased intracranial pressure will receive a lumbar puncture.
  Arms: Patients with increased intracranial hypertension
Diagnostic Test: Optical Coherence Tomography (OCT) imaging — Optical Coherence Tomography (OCT) imaging will measure the peripapillary retinal nerve fiber layer (RNFL) thickness measurements The images with enhanced depth imaging will be obtained to measure the Bruch's membrane orientation.
Diagnostic Test: Optic nerve B-scan ultrasound — Ultrasound will be used to measure the optic nerve sheath diameter 3 mm posterior to the posterior scleral surface.

SUMMARY:
Investigators will compare magnetic resonance (MR) elastography measurements to other forms of noninvasive methods of detecting raised intracranial pressure, including optical coherence tomography (OCT) imaging measurements of the retinal nerve fiber layer (RNFL) and indirect signs of raised intracranial pressure on magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
The goal of this study is to evaluate the brain elasticity in patients with idiopathic intracranial hypertension (IIH) and other forms of raised intracranial pressure, such as obstructive hydrocephalus. Investigators will evaluate for a correlation between brain stiffness and opening pressure on lumbar puncture. Investigators will also evaluate for changes in brain stiffness after interventions that are aimed at lowering intracranial pressure, including lumbar punctures, medications, and surgical interventions, such as ventriculoperitoneal shunts. Lastly, investigators will compare MR elastography measurements to other forms of noninvasive methods of detecting raised intracranial pressure, including optical coherence tomography (OCT) measurements of the retinal nerve fiber layer (RNFL) and indirect signs of raised intracranial pressure on MRI.

ELIGIBILITY:
All subjects will have the following inclusion criteria:

* Group 1: Papilledema from idiopathic intracranial hypertension and other forms of elevated intracranial pressure, including obstructive hydrocephalus
* Group 2: Patients without raised intracranial pressure.

All subjects will have the following exclusion criteria:

* Age <18
* Pregnancy (self-reported)
* Individuals for whom MR is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-01-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
MR elastography measurement of the brain elasticity | 1-2 weeks prior to lumbar puncture
  The primary outcome measure is the difference in the brain elasticity on MR elastography between patients with raised intracranial pressure and those with normal intracranial pressure

SECONDARY OUTCOMES:
MRI finding | 1--2 weeks prior to lumbar puncture
  The secondary outcome measurement are the retinal nerve fiber layer (RNFL) thickness and Bruch's membrane configuration on the MRI findings of raised intracranial pressure (optic nerve sheath diameter and pituitary/sella ratio). The cutoff from abnormal-to-normal will be established. The sensitivity and specificities will be established and compared against the other secondary outcome measurements and against MR elastography.
Ocular Coherence Tomography (OCT) finding | 1--2 weeks prior to lumbar puncture
  The secondary outcome measurements are the retinal nerve fiber layer (RNFL) thickness and Bruch's membrane configuration using ocular coherence tomography (OCT) of raised intracranial pressure (optic nerve sheath diameter and pituitary/sella ratio). The cutoff from abnormal-to-normal will be established. The sensitivity and specificities will be established and compared against the other secondary outcome measurements and against MR elastography
Optic Nerve B-scan ultrasound finding | 1--2 weeks prior to lumbar puncture
  The secondary outcome measurement are the retinal nerve fiber layer (RNFL) thickness and Bruch's membrane configuration on the optic nerve B-scan ultrasound findings of raised intracranial pressure (optic nerve sheath diameter and pituitary/sella ratio). The cutoff from abnormal-to-normal will be established. The sensitivity and specificities will be established and compared against the other secondary outcome measurements and against MR elastography.

CONTACTS AND LOCATIONS:
Overall Officials: John J Chen, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials